CLINICAL TRIAL: NCT00888485
Title: Secondary Prevention in Uppsala Primary Health Care After Myocardial Infarction, Coronary Artery CABG and PCI. Secondary Prevention After CHD (SUPRIM).
Brief Title: Randomized Trial of Behavioral Intervention Versus Standard Treatment
Acronym: SUPRIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Professor Kurt Svärdsudd, Section head, Uppsala University, Department of Public Health and Caring Scienses
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SMRK97; Vardal V96; FAS F0196; SOS 1471; SHLA E010
Record Dates: First submitted 2009-04-24; First posted 2009-04-27 (Estimated); Last update posted 2009-04-27 (Estimated); Status verified 2009-04

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral intervention (Experimental): Group exposed to behavioral intervention program
  Interventions: Behavioral: Behavioral interventional program
- Standard treatment (Active Comparator)
  Interventions: Behavioral: Behavioral interventional program

INTERVENTIONS:
Behavioral: Behavioral interventional program — Cognitive behavioral therapy intervention adapted to coronary disease patients performed in 20 group sessions during one year.

SUMMARY:
The purpose of this study is to determine the possible preventive effect of behavioural modification versus standard treatment after hospital discharge in CHD patients.

DETAILED DESCRIPTION:
According to a recent Cochrane report there is little evidence so far that psychological interventions affected total or cardiac mortality, but had a reduction in the number of non-fatal recurrent AMI and small effect on anxiety and depression.

The subjects were recruited among consecutive patients discharged from Uppsala University Hospital. Inclusion criteria were age 75 years or younger, discharged from the hospital after a myocardial infarction (AMI) or percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), living in the hospital primary catchment area, referred back to the general practitioner (GP) within one year after the hospital admission, not having previously participated in similar programs, being Swedish speaking, being willing to participate in the study, and accepting the random group allocation to be. All subjects fulfilling the inclusion criteria were informed about the study during the first outpatient visit to the hospital two weeks after discharge. During a visit to the cardiology outpatient department three months after discharge the informed subjects were formally invited to participate and verbal informed consent was obtained, standard requirement at the time. A written invitation letter to a baseline examination in the study was then mailed to the subjects and those who accepted the invitation were eventually included. The recruitment period lasted from may 1996 to august 2001 and the follow-up data collection was completed in 2008.

At the end of the recruitment period 812 consecutive patients had been considered for inclusion, of which 302 did not fulfill the inclusion criteria, and 148 subjects declined to participate, in most cases because of long distance from home to the hospital or lack of time. The remaining 362 subjects (71.0% of eligible cases), 85 (23%) women, 277 (77%) men gave informed consent to participation, of whom 185 (51.1%) had been admitted for an AMI, 122 (33.7%) for a CABG, and 55 (15.2%) for a PCI. Seventy-one AMI subjects had a PCI performed during the course of events and three had a CABG. At the time of the study more than 95% of the Swedish population in these age groups was Caucasians and about 90% were native Swedes.

The group allocation was based on the SAS "ranuni" function that provides random numbers with equal probability. The randomization procedure was based on pre-prepared sealed envelopes with a serial number on the outside and containing a paper sheet with the group allocation on the front side and a blinding print on the back to eliminate the possibility to read the group allocation sheet from the outside of the envelope. The envelopes were kept in sorted ascending serial number order in a safe. After inclusion of a subject the study monitor (the only person with access to the randomization envelopes and information) drew the next envelope in order and inserted the allocation paper sheet in the study protocol. Of those included, 192 were allocated to behavioral intervention and 170 to the reference group. The included subjects were informed about the group allocation after the baseline measurement.The subjects received an invitation letter for a first (baseline) examination and a first postal questionnaire. The procedure was repeated at the 6th, 12th, 18th and 24th month after baseline. The examination included anthropometry (height, weight and sagittal diameter), and blood pressure measurement, and blood sampling for blood lipids.

Information on marital status, educational level, smoking habits, job status (including retirement or on sick leave), social background and lifestyle factors was obtained by questionnaire.

The Gothenburg Quality of Life Instrument, previously validated and used in many studies, was used to measure quality-of-life aspects. Information on medical history until the baseline measurement was obtained from the baseline questionnaire. The subjects were asked whether they had experienced angina pectoris, hypertension, hyperlipemia, congestive heart failure, stroke, peripheral artery disease, diabetes, or asthma/congestive pulmonary disease. Responses were given as "yes" or "no".

Hospital admission data were obtained by linking the study data set to the National Hospital Discharge Register and the National Cause of Death Register to include non-fatal as well as fatal events. The record linkage was based on the unique personal identification number (PIN) given to all Swedish residents at birth or immigration and used in all official registers, including the population register. The PIN is based on year, month and day of birth, and a four-digit serial number. The second last serial number digit refers to subject sex and the last digit is a control digit, by which the correctness of the PIN easily can be checked and if necessary corrected against the population register. Data from the National Hospital Discharge Register included all hospital admissions from 1971 until 31 December 2006.

Survival data were obtained from the Cause of Death Registry, including all deaths in the study population until 31 December 2006. The overall autopsy rate was 23%, and the autopsy rate among those who had a first fatal cardiovascular event as outcome in the trial was 50%.

Diagnoses in the Hospital Discharge Register and the Cause of Death Register were coded according to the International Classification of Diseases (ICD). Cardiovascular disease was defined as ICD-8 codes (until 1986) and ICD-9 codes (1987-1996) 401-459, and ICD-10 codes (from 1997 on) I00-I99. Acute myocardial infarction was defined as ICD-8 code 410, ICD-9 code 410, and ICD-10 code I21-I22.

Based on these data the number of AMIs per subject prior to baseline was identified. In addition, all death irrespective of its cause, first cardiovascular disease event, fatal or non-fatal was identified, as well as the first AMI post baseline.

Subjects entered the intervention program within a year after the index coronary event. The intervention was based on cognitive behavioral therapy focused on stress management aimed to help CHD patients cope with stress and reduce experience of daily stress, time deadlines and hostility. For this purpose they were randomized to behavioral intervention or no behavioral intervention (usual care). The intervention, cognitive behavioral therapy (CBT), adapted to CHD patients, was performed in group-sessions, including 5-8 participants, separate groups for women and men, altogether 20 two-hour sessions per group during one year. An experienced psychologist, expert in CHD patient CBT, formed a team of trained psychologists and nurses, and together they performed the sessions. To secure continuity, all groups were treated by the same group leader. Attendance rate in sessions was monitored and the adherence to the program was excellent. Median attendance rate was 85%, and less than 5% attended less than 50% of the sessions. The program had specific goals and 5 key components; education, self-monitoring, skills training, cognitive restructuring and spiritual development.

ELIGIBILITY:
Inclusion Criteria:

* Discharged from hospital with CHD
* Age 75 years or less
* Living in hospital catchment area
* Able to understand Swedish
* Willing to accept randomized group

Exclusion Criteria:

* Psychiatric disease
* Participated in similar study previously

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 1996-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Admission to hospital for recurrent CHD event | 8 years

SECONDARY OUTCOMES:
Quality of life measures | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Svärdsudd, MD PhD, Principal Investigator — Uppsala University

REFERENCES:
- [Result] Gulliksson M, Burell G, Lundin L, Toss H, Svardsudd K. Psychosocial factors during the first year after a coronary heart disease event in cases and referents. Secondary Prevention in Uppsala Primary Health Care Project (SUPRIM). BMC Cardiovasc Disord. 2007 Nov 21;7:36. doi: 10.1186/1471-2261-7-36. PMID 18031575
- [Derived] Gulliksson M, Burell G, Vessby B, Lundin L, Toss H, Svardsudd K. Randomized controlled trial of cognitive behavioral therapy vs standard treatment to prevent recurrent cardiovascular events in patients with coronary heart disease: Secondary Prevention in Uppsala Primary Health Care project (SUPRIM). Arch Intern Med. 2011 Jan 24;171(2):134-40. doi: 10.1001/archinternmed.2010.510. PMID 21263103